CLINICAL TRIAL: NCT02310464
Title: An Open-Label Study to Assess the Safety, Tolerability, and Efficacy of Active Immunotherapy With Dose Escalation and Cohort Expansion of OBI-833 (Globo H-CRM197) in Advanced/Metastatic Gastric, Lung, Colorectal, or Breast Cancer Subjects
Brief Title: Trial of Active Immunotherapy With OBI-833 (Globo H-CRM197) in Advanced/Metastatic Gastric, Lung, Colorectal or Breast Cancer Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OBI Pharma, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OBI-833-001
Record Dates: First submitted 2014-12-02; First posted 2014-12-08 (Estimated); Results first posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Metastatic Gastric Cancer; Metastatic Breast Cancer; Metastatic Colorectal Cancer; Metastatic Lung Cancer
MeSH Terms: conditions — Stomach Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Experimental): Each subject will be given a total of 10 doses of OBI-833/OBI-821 subcutaneously at weeks 1,2,3,4,6,8,12,16,20,and 24 (Visits 1,2,3,4,5,6,7,8,9 and 10, respectively). Post treatment, subjects will be continually evaluated for safety and immune response every 4 weeks until the end of study, which is 12 weeks after the last dose, i.e., week 36. Subsequently, subjects will be followed for survival every 8 weeks up to 12 months after the end of study.
  Interventions: Drug: OBI-833/OBI-821
- Cohort expansion phase (Experimental): Each subject will be given OBI-833/OBI-821 at Weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, and every 8 weeks thereafter (Visits 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, and every 8 weeks thereafter) until disease progression. For the subjects discontinued treatment because of disease progression, subjects will be continually evaluated for safety and immune response every 8 weeks until the end of the study, which is 24 weeks after the last dose.
  Interventions: Drug: OBI-833/OBI-821

INTERVENTIONS:
Drug: OBI-833/OBI-821

SUMMARY:
The purpose of this clinical study is to assess the safety and tolerability and efficacy of active immunotherapy with dose escalation and cohort expansion of OBI-833 in advanced/metastatic gastric, lung, colorectal, or breast cancer subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥21 years of age
2. Dose escalation phase: Histologically or cytologically confirmed diagnosis of gastric, lung, colorectal or breast cancer on file Cohort expansion phase: Histologically or cytologically confirmed diagnosis of Globo H-positive NSCLC
3. Dose escalation: Subjects with recurrent or metastatic incurable disease that failed to respond to at least one line of anticancer standard therapy and for which standard treatment is no longer effective or tolerable.

   Cohort expansion phase: Subjects with recurrent or metastatic NSCLC who have achieved stable disease (SD), or partial response (PR) status after at least 1 regimen of anticancer therapy (i.e., chemotherapy, or targeted therapy, or PD-1/PD-L1 antagonists either alone or in combination) , and there are no standard treatments available except permitted Target or PD-1/PD-L1 therapies
4. Measurable disease (i.e., present with at least one measurable lesion per RECIST, version 1.1.
5. Dose Escalation Phase: No known central nervous system (CNS) metastases or neurological symptoms possibly related to active CNS metastasis in Dose Escalation Phase.

   Cohort Expansion Phase: Subjects with asymptomatic CNS metastases for at least four weeks before study drug treatment
6. Performance status: ECOG ≤ 1
7. Organ Function Requirements - Subjects must have adequate organ functions as defined below:

   AST/ALT ≤ 3X ULN (upper limit of normal) AST/ALT ≤ 5X ULN [with underlying liver metastasis] Total bilirubin ≤ 2.0 X ULN Serum creatinine ≤ 1.5X ULN ANC ≥ 1500 /µL Platelets > 100,000/µL
8. Subjects of child-bearing potential must agree to use acceptable contraceptive methods during treatment and until the end of the study. Subject not of childbearing potential (i.e., permanently sterilized, postmenopausal) can be included in study. Postmenopausal is defined as 12 months with no menses without an alternative medical cause.
9. Ability to understand and the willingness to sign a written informed consent document according to institutional guidelines.

Exclusion Criteria:

1. Patients who have not received standard chemotherapy, hormonal or targeted therapy for their underlying advanced/metastatic cancer.
2. Subjects who are pregnant or breast-feeding at entry.
3. Subjects with splenectomy.
4. Subjects with known or clinically manifest, symptomatic CNS metastases in Dose Escalation Phase.
5. Subjects with HIV infection, active hepatitis B infection or active hepatitis C infection.
6. Subjects with any autoimmune disorders requiring iv/oral steroids or immunosuppressive or immunomodulatory therapies.

   - e.g., Type 1 juvenile onset diabetes mellitus, antibody positive for rheumatoid arthritis, Grave's disease, Hashimoto's thyroiditis, lupus, scleroderma, systemic vasculitis, hemolytic anemia, immune mediated thrombocytopenia, etc.
7. Subjects with any known uncontrolled inter-current illness including ongoing or active infections, symptomatic congestive heart failure (NYHA>2), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Dose escalation phase: Subjects with any of the following MEDICATIONS within 4 weeks prior to IP treatment, except permitted therapies as listed in section 7.1:

   * Chemotherapeutic Agent
   * Immunotherapy [mAbs, Interferons, Cytokines (except GCSF)]
   * Immunosuppressants (e.g., cyclosporin, rapamycin, tacrolimus, rituximab, alemtuzumab, natalizumab, etc.).
   * IV/oral steroids except single prophylactic use in CT/MRI scan or other one-time use in approved indications. The interval between IV/oral steroids administration and first dose of OBI-833/OBI-821 must be more than pharmacological duration or 5 half-lives of administered steroids, whichever is the longer. Uses of inhaled and topical use of steroids are allowed.
   * Another investigational drug

   Cohort Expansion Phase: Subjects with any of the following MEDICATIONS within 4 weeks prior to IP treatment, except permitted therapies:
   * Chemotherapeutic Agent
   * Immunotherapy [Interferons, Cytokines] (except PD-1/PD-L1 antagonists)
   * Immunosuppressants (e.g., cyclosporin, rapamycin, tacrolimus, rituximab, alemtuzumab, natalizumab, etc.).
   * IV/oral steroids except single prophylactic use in CT/MRI scan or other one-time use in approved indications. The interval between IV/oral steroids administration and first dose of OBI-833/OBI-821 must be more than pharmacological duration or 5 half-lives of administered steroids, whichever is longer. Uses of inhaled and topical steroids are allowed.
   * Another investigational drug
9. Subjects with pleural effusions and/or ascites, due to malignancy, requiring paracentesis every 2 weeks or more frequently.
10. Subjects with any known severe allergies (e.g., anaphylaxis) to any active or inactive ingredients in the study drugs.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2021-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Escalation - Cohort 1: 10 μg OBI-833/100 μg OBI-821
- Dose Escalation - Cohort 2: 30 μg OBI-833/100 μg OBI-821
- Dose Escalation - Cohort 3: 100 μg OBI-833/100 μg OBI-821
- Expansion Cohort: NSCLC patients receiving 30 μg OBI-833/100 μg OBI-821
Period: Overall Study
Arm/Group | Dose Escalation - Cohort 1 | Dose Escalation - Cohort 2 | Dose Escalation - Cohort 3 | Expansion Cohort
Started | 4 | 3 | 4 | 14
Completed | 0 | 0 | 0 | 1
Not Completed | 4 | 3 | 4 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation - Cohort 1 | Dose Escalation - Cohort 2 | Dose Escalation - Cohort 3 | Expansion Cohort | Total
Number analyzed (Participants) | 4 | 3 | 4 | 14 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3 | 11 | 17
  >=65 years | 3 | 1 | 1 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (10.61) | 65 (10.44) | 58 (9.42) | 59.2 (10.25) | 60.3 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 7 | 16
  Male | 1 | 0 | 1 | 7 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 4 | 14 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 14 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 2
  White | 3 | 2 | 2 | 0 | 7
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 0 | 9
  Taiwan | 1 | 0 | 1 | 14 | 16
Cancer Type [Count of Participants; unit: Participants]
  Colorectal | 3 | 1 | 4 | 0 | 8
  Lung | 1 | 0 | 0 | 14 | 15
  Breast | 0 | 2 | 0 | 0 | 2
Tumor Globo H Expression [Mean (Standard Deviation); unit: scores on a scale] — Tumor samples were tested for Globo H expression by immunohistochemistry (IHC). The % of tumor cells with complete/partial membrane and/or cytoplasmic Globo H expression were recorded at each staining intensity - 0 for no detectable stain; 1+ for translucent or low-level stain; 2+ for moderate or opaque stain; 3+ for strong or solid stain. The H-score values [0 (no expression) to 300 (full expression)] were calculated as follows:
  H-score = [(% of tumor cell membrane/cytoplasmic at 1+) x 1 + (% of tumor cell membrane/cytoplasmic at 2+) x 2 + (% of tumor cell membrane/cytoplasmic at 3+) x 3] Population: Subjects in the dose escalation phase were not screened for Globo H expression. Only subjects in the cohort expansion phase were screened for Globo H expression for enrollment.
  scores on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    (all) |  |  |  | 130.6 (83.77) | 130.6 (83.77)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Time Frame: Approximately 13 weeks for dose escalation cohorts and 44 weeks for expansion cohort
Measure: Number; unit: Participants
Arm/Group | Dose Escalation - Cohort 1 | Dose Escalation - Cohort 2 | Dose Escalation - Cohort 3 | Expansion Cohort
Number analyzed (Participants) | 4 | 3 | 4 | 14
Participants
  Serious TEAEs | 1 | 0 | 3 | 3
  Any TEAEs | 4 | 3 | 4 | 13

2. Secondary Outcome: Maximal Post-baseline Anti-Globo H Antibody Responses
Description: Anti-Globo H IgM and IgG concentrations were measured using a chemical binding assay.
Time Frame: Approximately 13 weeks for dose escalation cohorts and 44 weeks for expansion cohort
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Dose Escalation - Cohort 1 | Dose Escalation - Cohort 2 | Dose Escalation - Cohort 3 | Expansion Cohort
Number analyzed (Participants) | 4 | 3 | 4 | 14
μg/mL
  Maximal post-baseline anti-Globo H IgM concentration | 4.602 [0.392 to 54.081] | 2.048 [1.116 to 3.758] | 3.165 [2.322 to 4.315] | 13.920 [5.835 to 33.207]
  Maximal post-baseline anti-Globo H IgG concentration | 5.011 [0.209 to 120.156] | 1.000 [NA to NA] — All three subjects had the same maximal IgG concentration, i.e. no variation. Therefore, the CI (calculated using the variance) cannot be calculated, i.e. not available. | 2.186 [0.406 to 11.783] | 9.472 [4.372 to 20.523]

ADVERSE EVENTS:
Time Frame: Approximately 13 weeks for dose escalation cohorts and 44 weeks for expansion cohort.
Arm/Group | Dose Escalation - Cohort 1 | Dose Escalation - Cohort 2 | Dose Escalation - Cohort 3 | Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/3 | 1/4 | 3/14
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 3/4 | 3/14
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 4/4 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation - Cohort 1 (N=4) | Dose Escalation - Cohort 2 (N=3) | Dose Escalation - Cohort 3 (N=4) | Expansion Cohort (N=14)
Disease Progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation - Cohort 1 (N=4) | Dose Escalation - Cohort 2 (N=3) | Dose Escalation - Cohort 3 (N=4) | Expansion Cohort (N=14)
Injection site induration (General disorders) | 3 (7) | 3 (8) | 2 (5) | 0 (0)
Injection site erythema (General disorders) | 2 (10) | 3 (14) | 2 (4) | 0 (0)
Injection site pain (General disorders) | 1 (6) | 3 (17) | 2 (12) | 1 (4)
Injection site pruritus (General disorders) | 1 (1) | 1 (2) | 1 (6) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 2 (3) | 1 (6) | 7 (35)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Injection site paraesthesia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (3)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (14)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RBC sedimentation rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device occlusion (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Burning sensations (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivaloedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT02310464/Prot_000.pdf